CLINICAL TRIAL: NCT03039010
Title: Validation of Data for Dental Health in the SKaPa Registry for Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Tita Mensah (Other)
Responsible Party: Sponsor-Investigator, Tita Mensah, Paediatric dentist, PhD candidate, Malmö University
Organization: Malmö University (Other)
Other Study IDs: MalmoU
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Swedish Quality Registry for dental health care (SKaPa) is a national registry that has since year 2008 gathered dental data. The data is automatically extracted from the patients' electronical dental data records. A vast majority of the public dental health care clinics deliver data on a daily basis (SKaPa, 2013). SKaPa has the purpose to improve and develop the quality of care and patient outcomes for both prevention and reparative/restorative methods concerning caries and periodontal disease. For children and adolescents, it is above all information related to dental caries that is collected (SKaPa, 2013). So far, SKaPa has published seven annual reports. In the report for year 2013 a limited information about the status of children was given, due to uncertainty in the quality of the information that is passed on to SKaPa (SKaPa, 2013). There is therefore a need to examine the validity of the data supplied to SKaPa.

Tooth decay is the most common disease in children and adolescents that often lead to invasive interventions and pain. There are reports of great social disparities in dental health in children and adolescents in Sweden (The National Board of Health and Welfare, Socialstyrelsen, 2013). Because tooth decay is a common disease in children, it is important to be able to monitor the occurrence of the disease and also examine how it differs across various groups of children and adolescents. This is now possible through the several registries that are available in the dental and health care. Register-based research will be an important tool to ensure that children and adolescents receive oral health and dental care on the same premise as others, provided the data in the registries are valid. Furthermore, register-based research is important for development and quality assurance of dental care.

DETAILED DESCRIPTION:
Validation of data for dental health in the SKaPa registry for children and adolescents.

Research question: How reliable is the information on dental caries of children and adolescents in the SKaPa registry?

Hypothesis: Data to SKaPa differences minimally compared with medical records and clinical status when it comes to deft/DMFT for 6 and 12 year old children. There is an underregistration of dental caries due to not registering caries that will not be treated. The children that are examined with bite-wings will have a higher score of deft/DMFT than other children.

Method: Tooth decay is examined clinically by trained and calibrated dentists in 170 6-year-olds and12-year-olds will be included. The registrations are compared with the most recently collected data for individuals in SKaPa to evaluate the quality of the information in the SKaPa registry. The inclusion of patients for the clinical dental examinations is based on cluster sampling (dental clinic in the Public Dental Service) in Värmland. The exact number of individuals being examined is determined after power calculation in collaboration with a Biostatistician.

Furthermore, a randomized sample of 500 individuals where data reported to SKaPa for the year 2014 will included for evaluation of dental records and dental radiographs. Comparisons are made between the data in the registry with the original data in the patient record. Preliminary calculated 250 6-year-olds and 250 12-year-olds will be included. Study population size is determined after power-calculation and in collaboration with a statistician. The study would make it possible to detect differences in deft/DMFT at 10% with a standard deviation of 30%. The reviews of the dental records are made by two calibrated dentists. The consistency of registrations from dental records and radiographs are continually evaluated throughout study. Primary outcome measures in both the clinical part and the dental record survey are number of teeth and deft/ DMFT.

The following data are registered:

* Status: Number of teeth, which teeth, manifest caries
* Radiographs - manifest caries lesions, and quality of radiographs - for example; possi-bility to see all interdental spaces, overlaps, marginal bone, quality of radiographic exposure
* Recordings in the dental records about patient's health status, medications, risk assessment
* Therapy decisions about diagnosed manifest tooth decay
* Undiagnosed manifest caries
* Prevention treatments
* Which dental profession the child has met (dentist/dental hygienist/dental assistant)
* Decision about when the next examination is planned
* When the previous examination was done, was X-rays taken (yes/no), diagnosed caries initially/manifest/or not

ELIGIBILITY:
Inclusion Criteria:

* The inclusion of patients for the clinical dental examinations is based on cluster sampling (dental clinic in the Public Dental Service) in Värmland.

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Study part 1: A total of 170 individuals (6-year-olds and 12-year-olds) will be included.
  Part 2: A total of 500 individuals patient journals.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Number of teeth and deft/ DMFT | 10 minutes
  The dental caries index DMFT is commonly used to measure caries prevalence. DMFT means Decayed, Missing, Filled Teeth, i.e. carious, missing (due to tooth decay) and filled teeth in permanent dentition. In the primary dentition the terms used are; d (decayed), e (extracted) and f (filled) teeth.

CONTACTS AND LOCATIONS:
Locations (1):
- National dental Service, Folktandvården Värmland, Karlstad, Värmland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mensah T, Tranaeus S, Cederlund A, Naimi-Akbar A, Klingberg G. Swedish quality registry for caries and periodontal diseases (SKaPa): validation of data on dental caries in 6- and 12-year-old children. BMC Oral Health. 2021 Jul 24;21(1):373. doi: 10.1186/s12903-021-01705-x. PMID 34301237